CLINICAL TRIAL: NCT02752711
Title: Validation of the PECARN Clinical Decision Rule for Children With Minor Head Trauma: a French Multicenter Prospective Study
Brief Title: Validation of the PECARN Clinical Decision Rule for Children With Minor Head Trauma
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0111
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Head Injury
Keywords: Minor head trauma; Children; Clinical decision rule
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: the PECARN clinical decision rule — the PECARN clinical decision rule for the detection of clinically-important traumatic brain injuries in children with minor head trauma

SUMMARY:
To date, the Pediatric Emergency Care Applied Research Network (PECARN) rule for identifying children who are at very low risk of clinically-important traumatic brain injuries after minor head trauma has not been validated prospectively in an independent population. Our goal was to evaluate the diagnostic performance of the PECARN clinical decision rule in a French pediatric population in multiple clinical settings.

DETAILED DESCRIPTION:
Head injury is a frequent reason for consultation with pediatric emergencies, over 95% are mild head injury defined by a Glasgow score greater than or equal to 13. In October 2009, the Pediatric Emergency Care Applied Research Network has published a rule clinical decision support of mild head injury of the child with the aim to identify children at very low risk for clinically severe intracranial lesions in order to avoid the use of CT and unnecessary exposure to radiation ionizing. This clinical decision rule constructed from a multicenter prospective cohort 42,412 American children allows on anamnestic and clinical elements to guide medical decision for conducting brain imaging, hospital monitoring or discharge home placing the child in three levels of risk of clinically severe intracranial lesions.

Since March 2012, the French Emergency Medicine Society recommends for the treatment of mild head trauma the child's use of the clinical decision rule provided that it is the subject of a validation study externally. Indeed, after the construction phase and before its daily application, a clinical decision rule must be subject to an broad validation process so that its predictive performance can be definitively established.

The investigators' work aims to conduct this broad validation study prospective multicenter way in a French pediatric population, as recommended by the French Emergency Medicine Society, in order to confirm or deny its predictive performance and allow its application and generalization. The investigators will check and if the clinical decision rule is adapted or not to the management of mild head injuries in the French pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children under 16 years admitted to an emergency room for mild head injury (Glasgow Coma Scale score ≥14) in the previous 24 hours
* Children who have agreed to participate in the study (if age> 8 years)
* Patient Parents have accepted the participation of their child in the study

Exclusion Criteria:

* Children with bleeding disorders
* Ventricular shunt Presence
* Benin mechanism of trauma (fall of the height of the child or impact against an object while walking / running with no sign that the scalp dermabrasion)
* Penetrating trauma
* Known brain tumor
* Previously known neurological disorders
* Evaluation scanographic in another hospital before emergency review

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In the study we included all children under 16 years of age admitted to the emergency room with mild head trauma with a Glasgow score greater than or equal to 14, occurred in the previous 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 1499 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically severe intracranial injury and classified at risk (top and middle) according to clinical decision rule in all patients with severe intracranial lesions | one month

CONTACTS AND LOCATIONS:
Overall Officials: Fleur LORTON, MD, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - Departmental Hospital of Vendée, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - Hospital of Saint-Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Derived] Lorton F, Poullaouec C, Legallais E, Simon-Pimmel J, Chene MA, Leroy H, Roy M, Launay E, Gras-Le Guen C. Validation of the PECARN clinical decision rule for children with minor head trauma: a French multicenter prospective study. Scand J Trauma Resusc Emerg Med. 2016 Aug 4;24:98. doi: 10.1186/s13049-016-0287-3. PMID 27488722